CLINICAL TRIAL: NCT02539017
Title: The Clinical Significance of Cellular Immune Adjuvant Therapy of Triple Negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: because of safety problem, this trial was stopped in the hospital
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renyu-012
Record Dates: First submitted 2015-08-05; First posted 2015-09-02 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: cellular immune therapy; triple negative breast cancer; adjuvant therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy; Immunotherapy

ARMS (2):
- Combined (Experimental): Combined Chemo Therapy and immunotherapy with double dendritic cell (DC) and cytokine-induced killer (CIK) cell
  Interventions: Drug: Chemo; Biological: Immunotherapy
- Chemo (Active Comparator): Control group: Chemo Therapy group
  Interventions: Drug: Chemo

INTERVENTIONS:
Drug: Chemo — Epirubicin,75mg/m2,intravenous ,on day 1 of each 21 day cycle, 4 cycles Cyclophosphamide,0.6g/m2,intravenous, on day 1 of each 21 day cycle, 4 cycles Docetaxel,75mg/m2, intravenous, on day 1 of each 21 day cycle, 4 cycles
Biological: Immunotherapy — Immunotherapy with double dendritic cell (DC)and cytokine-induced killer (CIK) cell
  Arms: Combined

SUMMARY:
As a special type of breast cancer, the triple negative breast cancer has the characteristics of high recurrence rate (2 years after surgery), high distant metastasis rate, poor prognosis and short survival time. No matter at home or abroad, the clinical researches of the triple negative breast cancer are mainly focused on finding new drugs and new treatment strategies in order to reduce its recurrence and distant metastasis rate. The DC/CIK cell immunotherapy combined with chemotherapy in the clinical study of metastatic triple negative breast cancer has already confirmed benefit. This study is based on the theory that the optimal timing of cellular immunity is while the host tumor load is under the smallest state. Put forward the hypothesis that the DC/CIK cell immunotherapy combined with chemotherapy may improve the disease-free survival and overall surviva after the triple negative breast cancer operation. The investigators intends to use the RCT, observing the clinical significance of cellular immune adjuvant therapy of triple negative breast cancer in 340 patients with TNBC. Do the safety evaluation of cellular immunity in the adjuvant treatment of breast cancer treatment, explore the clinical strategies for breast cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* ECOG score: ≤1
* the Primary invasive ductal carcinoma which are during the Ib period to IIIc and should be surgical resection while no distant metastasis (except for the tumor of N3 in the internal mammary region, the above clavicle LN), and the diagnosis of the tumor was confirmed by pathological diagnosis;
* There must be no residual in the surgical margin(except lobular carcinoma in situ), and the remove number of axillary lymph nodes in the same side must be above 10 (except for the negative sentinel lymph nodes).
* Have the results of the immunohistochemical detection of ER, PR and HER2, the one whose HER2+ and HER2++ should be confirmed by FISH.
* The chemotherapy regimens recommended by the guide and radiation therapy (qualified).
* Have normal tissue and organ function:

Bone marrow function: ANC must be≥1.5×109/L, the platelet count must be≥100×109/L , hemoglobin must be ≥10g/dL.

Renal function: serum creatinine must be≤1.5ULN Liver function: total bilirubin ≤1.5ULN，AST≤1.5ULN，ALT≤1.5ULN

* The results of imaging examination of the contralateral breast molybdenum, chest CT, abdominal B ultrasound and whole body bone scan should be required before the random.
* Sign the informed consent form.
* Have a good compliance, and can be follow-up for at least 5 years.

Exclusion Criteria:

* have the past history of breast cancer with the same or opposite side, a history of immune system diseases.
* T1aN0M0, inflammatory breast cancer and bilateral breast cancer; patients with T cell lymphoma.
* Have the history of other malignant tumors before (except for the cervical carcinoma in situ, squamous cell carcinoma of the skin, skin basal cell carcinoma).
* Have the important organ dysfunction of heart, lung, liver, kidney and others.
* People who are pregnant or unwilling to use contraception during treatment.
* Patients who have received organ transplantation or long-term use of immunosuppressive agents.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
disease free survival | up to 3 years

SECONDARY OUTCOMES:
overall survival | up to 3 years
percentage of participants with fever, skin rash, bone marrow suppression, allergy, gastrointestinal response, myalgia and arthralgia | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu Ren, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China